CLINICAL TRIAL: NCT00604994
Title: Prospective Evaluation of Lymphoedema Among Patients With Gynaecological Cancer
Acronym: LEGS
Status: Completed | Type: Observational
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: The University of Queensland (Other); Royal Brisbane and Women's Hospital (Other Government); Mater (Other); Mater Private Hospital (Other); Queensland Institute of Medical Research (Other); Queensland University of Technology (Other); Australia New Zealand Gynaecological Oncology Group (Other); Cancer Australia (Other)
Responsible Party: Sponsor
Other Study IDs: LEGS
Record Dates: First submitted 2008-01-13; First posted 2008-01-30 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Female Genital Diseases; Ovarian Cancer; Cervical Cancer; Endometrial Cancer; Vulval Cancer
Keywords: Lymphoedema; Gynaecology; Oncology; Malignant; Benign; Incidence
MeSH Terms: conditions — Genital Diseases, Female; Ovarian Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Vulvar Neoplasms; Lymphedema; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Malignant: Patients with malignant gynaecological conditions including cancers of the cervix, uterus, ovary, vulva and vagina
- Benign: Patients without malignant gynaecological cancers

SUMMARY:
This project will conduct a prospective, longitudinal, observational cohort study to assess the onset and incidence of lymphoedema, as well as investigate factors associated with its development among women newly diagnosed with gynaecological cancers in 2008 to 2011.

DETAILED DESCRIPTION:
Pathological swelling of the lower limbs (lymphoedema) is widely accepted to be a common consequence of treatment for gynaecological cancer. It is both a serious and debilitating complication, associated with significant morbidity, which impacts physically and emotionally on otherwise healthy women. Lymphoedema can also affect patients' ability to earn an income, especially if their work requires prolonged periods of standing or walking.

The causes of lymphoedema are largely unknown with clinical data scarce regarding its onset time and incidence after gynaecological cancer treatment.

The following hypotheses will be tested to address the aims of the project:

1. At least 20% of patients will develop lower-limb lymphoedema following gynaecological cancer treatment.
2. Patient's age, as well as their body mass index (BMI), area of residence, degree of physical exercise, type of disease (uterine, cervical, ovarian, vulval/vaginal cancer; benign disease), mode of treatment (extent of lymph node dissection, radiotherapy, chemoradiation) and delay in wound healing are independent risk factors for lower-limb lymphoedema.
3. Patients who develop lymphoedema after gynaecological cancer treatment, will experience increased pain, lower quality of life (including worse body-image), and decreased sexual & financial well-being, compared to those who do not develop lymphoedema.
4. There will be at least 10% difference in the incidence of lower-limb lymphoedema between patients treated for gynaecological cancer compared to benign diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for surgery of benign or malignant gynaecological diseases as determined jointly by the surgeon and the patient.
* Non-pregnant female patients.
* Over 18 years of age at time of surgery.
* Patients who understand the conditions of the study and are willing to participate for the length of the prescribed term of follow-up.
* Patients who are capable of, and have given, informed consent to their participation in the study.

Exclusion Criteria:

* Patients with a pacemaker.
* Allergies against adhesive electrodes and extensive internal metal plates are ineligible for BIS measurement.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with gynaecological conditons requiring treatment
Sampling Method: Non-Probability Sample
Enrollment: 761 (Actual)
Dates: Start 2008-06; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Time of onset of lymphoedema after gynaecological cancer treatment. | 2 years
Incidence of lymphoedema after gynaecological cancer treatment. | 2 years
Point prevalence of lymphoedema after gynaecological cancer treatment. | 2 years
Severity of lymphoedema after gynaecological cancer treatment. | 2 years

SECONDARY OUTCOMES:
Prevalence of key risk factors of post-treatment lymphoedema among patients with gynaecological cancer. | 2 years
Impact of risk factors on development of lymphoedema. | 2 years
Lymphoedema development in patients treated for gynaecological cancer compared to patients with benign disease. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Obermair, MD FRANZCOG CGO, Principal Investigator — Queensland Centre for Gynaecological Cancer
Locations (6):
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Wesley Hospital, Auchenflower, Queensland
  - Greenslopes Private Hospital, Greenslopes, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Mater Health Services, South Brisbane, Queensland
  - Royal Women's Hospital, Carlton, Victoria

REFERENCES:
- See also: QCGC Research — http://www.gyncan.org/